CLINICAL TRIAL: NCT07179003
Title: A Phase 2 Study of Methylene Blue Photodynamic Therapy for Treatment of Breast Abscesses
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Timothy Baran, Assistant Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00010960
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Breast Abscess
Keywords: Breast abscess; Drainage; Photodynamic therapy; Methylene blue
MeSH Terms: interventions — Methylene Blue; Fat Emulsions, Intravenous; Photochemotherapy

STUDY DESIGN:
Intervention Model Description: The study includes two arms: (1) standard of care breast abscess drainage and (2) MB-PDT plus standard of care breast abscess drainage.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MB-PDT + standard of care (Experimental): Each subject in this arm will receive standard of care breast abscess drainage, methylene blue, lipid emulsion, and laser illumination.
  Interventions: Procedure: Standard of care breast abscess drainage; Drug: Methylene Blue; Drug: Lipid Emulsion; Device: Insertion of optical fiber; Device: Laser illumination; Procedure: Photodynamic therapy
- Standard of care (Other): Each subject in this arm will receive standard of care abscess drainage
  Interventions: Procedure: Standard of care breast abscess drainage

INTERVENTIONS:
Procedure: Standard of care breast abscess drainage — All subjects will receive ultrasound-guided percutaneous abscess drainage in a procedure room. The site will be prepared and dressed following standard of care sterile procedure, and a needle/catheter will be advanced under ultrasound guidance into the abscess. The abscess will be drained by syringe aspiration, and the cavity will be flushed with sterile saline. Aspirated abscess fluid will be delivered to the Clinical Microbiology Laboratory for processing, including bacterial identification and antibiotic susceptibility testing.
Drug: Methylene Blue — Following standard of care breast abscess drainage, for subjects randomized to the photodynamic therapy arm, sterile, clinical-grade methylene blue will be infused into the abscess cavity at a concentration of 100 µg/mL via the same needle/catheter used for drainage. The volume introduced will be matched to the amount of abscess material aspirated during the standard of care drainage. After a 10-minute incubation interval, methylene blue will be aspirated and the cavity flushed with sterile saline to remove methylene blue that has not been taken up by microbes.
  Arms: MB-PDT + standard of care
Drug: Lipid Emulsion — For subjects randomized to the photodynamic therapy arm, immediately prior to illumination a lipid emulsion will be administered directly to the abscess through the drainage needle/catheter at a concentration of 0.1%. This lipid emulsion will be either Intralipid or Nutrilipid. The lipid emulsion serves to gently distend the cavity, and through light scattering, homogenize the light dose to the walls of the cavity. The volume administered will be matched to the amount of abscess material aspirated during the standard of care drainage. Following laser illumination, the lipid emulsion will be aspirated and the cavity flushed with sterile saline.
  Arms: MB-PDT + standard of care
Device: Insertion of optical fiber — For subjects randomized to the photodynamic therapy arm, a sterile, single-use optical fiber will be advanced to the approximate center of the abscess cavity via the same needle/catheter used for abscess drainage under ultrasound guidance. This will be connected to the clinical laser system via SMA connector for delivery of treatment light.
  Arms: MB-PDT + standard of care
Device: Laser illumination — For subjects randomized to the photodynamic therapy arm, laser illumination for photodynamic therapy will be delivered by a laser system operating at 665 nm (ML7710, Modulight, Tampere, Finland) at a fluence rate of 20 mW/cm^2. The laser power required to achieve this fluence rate will be calculated based on abscess size. Illumination will be delivered for ~20 minutes, resulting in a total delivered fluence of 25 J/cm^2.
  Arms: MB-PDT + standard of care
Procedure: Photodynamic therapy — For subjects randomized to the photodynamic therapy arm, the photodynamic therapy procedure comprises the methylene blue, lipid emulsion, insertion of optical fiber, and laser illumination interventions.
  Arms: MB-PDT + standard of care

SUMMARY:
The objective of this Phase 2 study is to evaluate the efficacy of methylene blue photodynamic therapy (MB-PDT) performed at the time of percutaneous breast abscess drainage for disinfection of breast abscesses. The study includes two arms: (1) standard of care breast abscess drainage and (2) MB-PDT plus standard of care breast abscess drainage. The primary endpoint is time to resolution of clinical symptoms. Secondary endpoints include imaging evidence of abscess resolution, abscess recurrence, need for repeated intervention, and cure rate across treatment groups. Responses will be compared between the two study arms for the per protocol population to determine the efficacy of MB-PDT relative to standard of care. The investigators hypothesize that the addition of MB-PDT to standard of care will significantly reduce the time to symptom resolution, compared to standard of care alone.

DETAILED DESCRIPTION:
Breast abscesses consist of a localized, walled-off collection of infected fluid within the breast, with symptoms including breast pain and inflammation, as well as nipple discharge, fever, chills, and nausea. If left untreated, breast abscesses can result in serious complications, including fistula formation and sepsis. The standard of care therefore involves draining the purulent fluid, generally under ultrasound guidance, and systemic antibiotic administration. Although this drainage procedure is typically technically successful, reported recurrence rates vary widely. These recurrent breast abscesses can require repeated drainage procedures, surgical intervention, extended hospital stays, and aggressive antibiotic regimens.

Photodynamic therapy (PDT), which relies upon the combination of photosensitive dyes known as photosensitizers, excitation by visible light, and molecular oxygen to generate bactericidal reactive oxygen species, represents a potentially powerful adjunct to standard of care drainage. The investigators have successfully completed a Phase 1 clinical trial assessing the safety and feasibility of methylene blue (MB) PDT at the time of percutaneous intra-abdominal abscess drainage. No adverse or serious adverse events were observed, and the procedure was well tolerated by all subjects. Based on the success of this Phase 1 clinical trial, the current study aims to assess efficacy of MB-PDT at the time of breast abscess drainage.

The investigators propose a randomized, controlled Phase 2 clinical trial, which will be conducted in accordance with the principles of good clinical practice and with approval by both the FDA and local IRB. Patients who have been diagnosed with a drainable abscess, that meet all inclusion/exclusion criteria, and have the approval of their primary care team, will be offered enrollment in the study at initial presentation. Consented subjects will be prospectively randomized using block randomization to one of two arms: (1) standard of care (SOC) percutaneous drainage and antibiotics alone or (2) PDT + SOC. The primary outcome is time to resolution of clinical symptoms. The secondary outcome is imaging evidence of abscess resolution, based on ultrasound tomography. Tertiary outcomes include abscess recurrence, need for repeated intervention, and cure rate across treatment groups.

The study population will consist of 50 subjects, allocated equally between the two groups. Sample size calculations are based on a hypothesized reduction in the time to resolution of clinical symptoms. The investigators use retrospective data from patients that received SOC at our institution over the course of 15 years to represent SOC, and the 18 subjects treated in our Phase 1 clinical trial in abdominopelvic abscesses to represent PDT. Retrospective standard of care patients had median time to resolution of 16 days (95% CI 14-18 days), while subjects treated with MB-PDT had a median time to resolution of 7 days (95% CI 3-14 days). This corresponds to a hazard ratio for resolution of symptoms of 3.5. The investigators target 90% power at a more conservative hazard ratio of 3.0 to determine the sample size in each arm. A sample size of 25 subjects per arm provides 90% power to detect a hazard ratio of 3.0 at a two-sided alpha=0.05 level of significance. With equal allocation between groups, this results in a total sample size of 50 participants, given that the investigators assume to fully observe the primary outcome in all subjects.

All subjects will receive standard of care ultrasound-guided percutaneous breast abscess drainage. The site will be prepared and dressed following standard of care sterile procedure, and a needle will be advanced under ultrasound guidance into the abscess. The abscess will be drained by syringe aspiration, and the cavity will be flushed with sterile saline. Aspirated abscess fluid will be delivered to the Clinical Microbiology Laboratory for processing.

For subjects randomized to the PDT arm, sterile methylene blue (MB) will then be administered to the abscess cavity using the same needle/catheter utilized for standard of care drainage. After a 10-minute incubation interval, MB will be aspirated and the cavity flushed with sterile saline. The abscess cavity will then be filled with sterile 0.1% lipid emulsion to gently distend the cavity, and through light scattering, homogenize the light dose to the walls of the cavity. A sterile optical fiber will be advanced to the approximate center of the abscess cavity via the same catheter/needle used for standard of care under image guidance. The proximal end of the fiber will be coupled to the output of a clinical laser system emitting light at 665 nm. Laser power will be delivered to the cavity at a constant fluence rate of 20 mW/cm^2. The laser power required to obtain the desired fluence rate at the wall will be calculated based on the abscess size. Illumination will be delivered for ~20 minutes, resulting in a total delivered fluence of 25 J/cm^2.

Immediately after laser irradiation, the Intralipid solution will be aspirated and the cavity again flushed with sterile saline. SOC drainage will then be completed, including cleaning of the skin surface and wound dressing.

All subjects will receive ultrasound tomography of their affected breast using an FDA-approved ultrasound tomography system located at our institution. This will be performed immediately pre- and post-intervention (SOC or PDT+SOC), and at follow-up appointments. From these images, the investigators will first extract the abscess volume and viscosity of the infected fluid on pre-procedure imaging. At each timepoint, abscess volume, abscess wall stiffness and density, and surrounding breast tissue stiffness and density will be extracted from imaging data.

A Cox proportional hazards model will be used to model time to clinical symptom resolution. A 1-degree of freedom likelihood ratio test comparing time to resolution between the control group (SOC alone) and the PDT group (PDT+SOC) will be used for the primary analysis. Abscess recurrence and need for repeated intervention will be compared between treatment groups using a Cox proportional hazards model. Cure rate will be compared between groups using Fisher's exact test. Imaging outcomes (breast abscess volume, density, stiffness) will be compared between groups using linear mixed-effects models, and will further be compared to radiologist measurements using Wilcoxon matched-pairs signed rank tests. Multivariable Cox proportional hazards models will be used to examine the effects of anatomical features, risk factors, and subject demographics on long-term treatment responses.

If successful, this research could demonstrate efficacy of PDT as an adjunct treatment for breast abscess patients that significantly reduces time to symptom resolution. The investigators hypothesize that this could also lead to reduced abscess recurrence. Ultimately, this would promote early recovery, reduce repeated intervention, and lead to lower overall health care costs for patients undergoing ultrasound-guided percutaneous breast abscess drainage.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years or older
* Clinical signs of breast abscess, including pain, redness, and/or heat of the breast
* Approval by the primary care team to pursue PDT and discuss enrollment with the patient

Exclusion Criteria:

* Pregnancy
* Lactation
* Allergy to contrast media, narcotics, sedatives, atropine or eggs
* Necrotic tissue that requires surgical debridement
* Severely compromised cardiopulmonary function or hemodynamic instability
* Thrombocytopenia (<50,000/mm3)
* Uncorrectable coagulopathy
* Poor kidney function (serum creatinine >3mg/dl)
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency
* Patients with hidradenitis suppurativa
* Patients with granulomatous mastitis
* Unable or unwilling to understand or to provide informed consent
* Unable or unwilling to undergo study procedures
* Patient unable to cooperate with, or to be positioned for the procedure
* Unable to comply with necessary follow up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2031-03 (Estimated); Study Completion 2031-03 (Estimated)

PRIMARY OUTCOMES:
Time to resolution of clinical symptoms | Day 1 post-intervention until resolution of symptoms
  Clinical symptoms will be scored daily using a standardized questionnaire that includes objective measures of fever, heart rate, and blood pressure, as well as subjective ratings of pain and heat of the breast using a Likert score. Time to resolution of clinical symptoms will be defined as the time from intervention to the first day on which subjects are afebrile and report no pain, redness, or heat of the breast.

SECONDARY OUTCOMES:
Abscess volume on ultrasound tomography | Day 14 post-intervention until resolution
  All subjects will receive ultrasound tomography of their breast immediately prior to abscess drainage, immediately following drainage, and at follow-up appointments. Follow-up imaging will occur at 14 days post-drainage, and every 14 days thereafter until abscess resolution. Images will be segmented to identify the abscess cavity and measure its volume in mL.

OTHER OUTCOMES:
Time to abscess recurrence | 6 months post-intervention
  Each subject's electronic medical record will be reviewed at 6 months post-intervention to determine whether there was recurrence of the treated abscess. If there was recurrence, time to recurrence in days will also be recorded.
Time to repeated intervention | 6 months post-intervention
  Each subject's electronic medical record will be reviewed at 6 months post-intervention to determine whether additional procedures were required to manage the treated abscess. If repeated intervention was required, the time from study intervention to repeated intervention in days will also be recorded.
Rate of abscess cure | 6 months post-intervention
  Each subject's electronic medical record will be reviewed at 6 months post-intervention to determine whether there was recurrence of the treated abscess, whether additional procedures were required to manage the treated abscess, and whether clinical symptoms resolved. If over this 6-month period there was no recurrence, no additional procedures were required to manage the abscess, and clinical symptoms resolved, this will be classified as a cure. If any of these conditions are not satisfied, this will be classified as not cured.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Rochester Medical Center, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No